CLINICAL TRIAL: NCT05842707
Title: Study of Cord Blood-derived CAR NK Cells Targeting CD19/CD70 in Refractory/Relapsed B-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aibin Liang，MD，Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Aibin Liang，MD，Ph.D., Director of Hematology and Oncology Center, Shanghai Tongji Hospital, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-008
Record Dates: First submitted 2023-03-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Refractory or Relapsed B-cell Non-Hodgkin Lymphoma
Keywords: B-cell Non-Hodgkin Lymphoma; CAR NK Cells Targeting CD19/CD70; Cord Blood-derived
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part 1 (dose escalation) and Part 2 (dose expansion) (Experimental): Part 1 (dose escalation)
  the dose of dualCAR-NK19/70 participants receive will depend on when you join this study. Up to 3 dose levels of dualCAR-NK19/70 will be tested. About 3-6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level of dualCAR-NK19/70. Each new group will receive a higher dose of dualCAR-NK19/70 than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of dualCAR-NK19/70 is found.
  Part 2 (dose expansion)
  Participants will receive dualCAR-NK19/70 at the recommended dose that was found in Part 1.
  Interventions: Drug: dualCAR-NK19/70 cell

INTERVENTIONS:
Drug: dualCAR-NK19/70 cell — Given by IV (vein)
  Other Names: CAR-NK cell

SUMMARY:
To find the highest tolerable dose of dualCAR-NK19/70 (a type of cell therapy) that can be given to patients who have B-cell lymphoma that is relapsed or refractory.

DETAILED DESCRIPTION:
Primary Objectives:

--The primary objective is to determine the safety and identify the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of dualCAR-NK19/70 in patients with r/r B-cell lymphomas.

Hypothesis: DualCAR-NK19/70 will be safe, well-tolerated, and effective in patients with r/r B-cell lymphomas.

Secondary Objectives:

--The secondary objective is to determine the efficacy in adults with r/r LBCL and FL grade 3B treated at the MTD or RP2D of dualCAR-NK19/70. Although the clinical benefit of dualCAR-NK19/70 has not yet been established, the intent of offering this treatment is to provide a possible therapeutic benefit, and thus the patient will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability. Secondary endpoints include overall response rate (ORR; including CR + PR) and CR rate as defined by the Lugano Classification response criteria for malignant lymphoma, DOR, PFS, and OS.

Exploratory Objectives:

--The exploratory objectives are to assess the cellular kinetics and pharmacodynamic effects of dualCAR-NK19/70 and to evaluate biomarkers associated with response, resistance, and toxicity after administration of dualCAR-NK19/70 in blood and tumor samples.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and sign the informed consent;
2. Age 18-75, male and female;
3. Histologically confirmed diffuse large B-cell lymphoma (DLBCL), transformed follicular lymphoma (tFL), primary mediastinal B-cell lymphoma (PMBCL), mantle cell lymphoma (MCL), and other Indolent B-cell NHL transforming types:

   （A） Relapsed or Refractory DLBCL and tFL after 2 lines Immunotherapy or chemotherapy ; （B） Definition of Refractory large B cell lymphoma (SCHOLAR - 1 Research Standard) : disease progression after more than 4 courses of standard Immunotherapy or chemotherapy; Or the time of disease stabilization ≤ 6 months; Or disease progression or recurrence within 12 months after autologous hematopoietic stem cell transplantation (auto-HSCT); （C） Relapsed or Refractory MCL must be 1 line with immune chemotherapy; BTK inhibitors are resistant or intolerant as 2-line therapy; （D） Relapsed or Refractory disease after chemotherapy including rituximab and anthracycline.
4. There was at least one measurable lesion with the longest diameter ≥ 1.5cm;
5. Estimated life expectancy of more than 12 weeks other than primary disease;
6. Previously confirmed diagnosis as CD19+ or CD70+ B-NHL.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 3.
8. Adequate reserve of organ function:

   （A） Serum alanine aminotransferase (ALT) / aspartate aminotransferase (AST) ≤2.5 times the Upper Limit of Normal (ULN) for age; （B） A creatinine clearance (as estimated either by a direct urine collection or Cockcroft-Gault Equation) > 60mL/min; （C） Total bilirubin and alkaline phosphatase ≤1.5 times the Upper Limit of Normal (ULN) for age; （D） glomerular filtration rate > 50 ml/min （E） Cardiac ejection fraction (EF) ≥ 45% as determined by an echocardiogram (ECHO) or Multigated Radionuclide Angiography (MUGA); （F） Baseline oxygen saturation >92% on room air （G） Absolute neutrophil count > 1000/μL, Platelet count > 45,000/μL ,Hemoglobin > 80g/L;
9. Once previous autologous hematopoietic stem cell transplantation (auto-HSCT) is allowed;
10. For systemic therapy(Such as systemic chemotherapy, systemic radiotherapy and immunotherapy), at least 3 weeks，for Targeted drug therapy alone，at least 2 weeks，must have elapsed at the time of cell infusion;
11. Either having failed or Relapsed after CAR-T therapy at 3 months of assessment;
12. Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study until the follow-up period of the study. Women of childbearing potential must have a negative serum or urine pregnancy test.
13. The viral load of severe coronavirus disease 2019 (COVID-19) is undetectable per quantitative PCR and/or nucleic acid testing for two tests.

Exclusion Criteria:

1. Allergic to any of the components of cell products;
2. Previous or concurrent of other type of maligant tumors;
3. Acute GvHD or generalized chronic GvHD with grade II-IV (Glucksberg standard) after previous autologous hematopoietic stem cell transplantation (auto-HSCT); Or receiving of anti-GVHD therapy;
4. Known history of systemic gene therapy within the prior 3 months;
5. Active systemic fungal, viral, or bacterial infection (except for simple urinary tract infections and bacterial pharyngitis), however, Preventive treatment is permitted;
6. Known history of infection with hepatitis B (HBsAg positive, but HBV-DNA<1000 is not excluded) or hepatitis C virus (including virus carriers), syphilis and other acquired and congenital immunodeficiency diseases, including but not limited to HIV infection;
7. Class III or IV heart failure as defined by the New York Heart Association;
8. Persisting toxicities (>grade 1, except for clinically non-significant toxicities such as alopecia, fatigue, and anorexia) due to prior trerapy;
9. Known history of active seizures or presence of seizure activities or other central nervous system disease;
10. Have evidence of central nervous system lymphoma(CNS lymphoma) on CT or MRI;
11. Breast-feeding woman;
12. Any circumstances that possibly increase the risk of subjects or interfere with study results, which judged by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2028-01-18 (Estimated); Study Completion 2029-01-18 (Estimated)

PRIMARY OUTCOMES:
incidence of dose limiting toxicity(DLTs) | up to 28 days
  To evaluate the safety,tolerabitility,and determine the recommended dosage of cord blood-derived CAR NK cells targeting CD19/CD70

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | 6 months
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70
Complete Remission Rate(CRR) | 3 months
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70
Overall survival(OS) | Up to 3 years
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70
Duration of Response(DOR) | Up to 3 years
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70
progression-free survival(PFS) | Up to 3 years
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70

OTHER OUTCOMES:
Incidence of Adverse Events | through study completion; an average of 1 year,up to 3 years
  Type, frequency, and severity of adverse events,Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5
Exploratory Objectives | Up to 3 years
  The exploratory objectives are to assess the cellular kinetics and pharmacodynamic effects of dualCAR-NK19/70 and to evaluate biomarkers associated with response, resistance, and toxicity after administration of dualCAR-NK19/70 in blood and tumor samples.

CONTACTS AND LOCATIONS:
Overall Officials: aibin Liang, Study Chair — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No